CLINICAL TRIAL: NCT03918707
Title: Utility of Rapid Whole Genome Sequencing in the NICU: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Illinois College of Medicine at Peoria (Other)
Collaborators: Rady Children's Institute of Genomic Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1346781
Record Dates: First submitted 2019-03-04; First posted 2019-04-17 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Genetic Disease; Genetic Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: The prospective group will consist of approximately 15 evaluable patients who will undergo rWGS sequencing in addition to standard of care genetic testing. Subjects in this study will be drawn from children admitted to the NICU at OSF HealthCare Children's Hospital of Illinois who meet inclusion criteria.
  Interventions: Diagnostic Test: Rapid Whole Genome Sequencing (rWGS)
- Historical Control: The historical control group will consist of patients admitted to the NICU between January 1, 2016 and December 31, 2018 who received genetic testing at less than 4 months of age and fulfil eligibility criteria.

INTERVENTIONS:
Diagnostic Test: Rapid Whole Genome Sequencing (rWGS) — rWGS will be performed on blood samples from subjects in the prospective group in addition to standard of care laboratory testing and imaging studies. Blood samples will also be obtained from biological parents (if available), to determine if variants are inherited or de novo and for variant segregation.
  Groups: Prospective

SUMMARY:
This is a pilot study involving a prospective group of 15 evaluable patients who will undergo rapid whole genome sequencing in addition to standard of care testing. Subjects will be drawn from children admitted to the NICU at OSF Health Care Children's Hospital of Illinois who meet inclusion criteria. The aims of this study are to evaluate the turn-around time and cost of performing rapid whole genome sequencing (rWGS) compared to standard of care in the diagnosis of genetic disorders among critically ill infants in a regional children's hospital and to describe management outcomes of utilizing rWGS in acutely ill patients less than four months of age.

ELIGIBILITY:
Inclusion Criteria:

Patients in the NICU less than 4 months of age with complex medical presentation of unknown etiology, who have 2 or more of the following are eligible:

* critically ill* and/or organ dysfunction
* one or more major congenital anomalies
* dysmorphic features and/or abnormal growth parameters
* neurologic impairment (seizure, hypotonia, encephalopathy)
* cardiomyopathy
* features suggestive of a metabolic disorder (eg unexplained/persistent hypoglycemia or acidosis)

  * critically ill - cardiorespiratory insufficiency requiring ventilatory or cardiac support

Exclusion Criteria:

* previously confirmed specific genetic diagnosis (antenatal or postnatal)
* obvious clinical findings for a specific condition that could be tested by targeted gene analysis
* preterm less than 24 weeks post-menstrual age
* ward of the state
* parent/legal guardian refusal to give consent for participation in the study
* patient does not meet eligibility criteria

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a pilot study involving a prospective group of approximately 15 evaluable patients who will undergo rWGS sequencing in addition to standard of care genetic testing. Subjects in this study will be drawn from children admitted to the NICU at OSF HealthCare Children's Hospital of Illinois who meet inclusion criteria. Non English speaking patients and their families may also be approached for participation in the study. Data will also be collected from a historical control of similar patients hospitalized from January 1, 2016 - December 31, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Turnaround Time | Duration of individual patients hospital stay typically less than 60 days
  If normally distributed, we will use t test for univariate analysis, and linear regression models for multivariate analysis to assess the intervention effects. Otherwise, we will use Wilcoxon two-sample t test or robust linear regression models. For other categorical variables, we will use chi-square to compare the difference between the prospective and historical control groups. Stratified analysis will be performed in order to get insight into the relationships of the data.
  We will analyze data within intervention, and control group, respectively. Means and standard deviations will be reported for continuous variables, and percentage values, odds ratio, 95% confidence interval will be reported for categorical variables. The two-tailed p values are calculated for all tests, and p<0.05 will be considered a statistically significant result. SAS 9.4 will be used for data management and data analysis.
Cost of Hospitalization until Genetic Diagnosis | Duration of individual patients hospital stay typically less than 60 days
  If normally distributed, we will use t test for univariate analysis, and linear regression models for multivariate analysis to assess the intervention effects. Otherwise, we will use Wilcoxon two-sample t test or robust linear regression models. For other categorical variables, we will use chi-square to compare the difference between the prospective and historical control groups. Stratified analysis will be performed in order to get insight into the relationships of the data.
  We will analyze data within intervention, and control group, respectively. Means and standard deviations will be reported for continuous variables, and percentage values, odds ratio, 95% confidence interval will be reported for categorical variables. The two-tailed p values are calculated for all tests, and p<0.05 will be considered a statistically significant result. SAS 9.4 will be used for data management and data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Illinois, Peoria, Illinois, United States